CLINICAL TRIAL: NCT06608810
Title: Comparison of Efficacy in Pectoral Nerve Block Type II, Thoracic Paravertebral Block, and General Anesthesia Alone for Excision of Breast Fibroma: a Prospective Randomized Controlled Trial
Brief Title: The Application of Pectoral Nerve II(PECS II)block in Breast Fibroadenoma Resection Surgery
Acronym: PECS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Baogang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-MER-069
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Nerve Block; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comparison of efficacy in pectoral nerve block type II, thoracic paravertebral block, and general an (Other)
  Interventions: Drug: nerve block with 0.5% ropivacaine

INTERVENTIONS:
Drug: nerve block with 0.5% ropivacaine — General anesthesia tracheal intubation was used. Induction was performed with midazolam 0.05ml/kg, etomidate 0.3-0.4mg/kg, sufentanil 0.3μg/kg-0.4μg/kg, and rocuronium bromide 0.8mg/kg, and after sufficient oxygen and denitration, the tracheal tube was placed by visual laryngoscopy, and the position of the tube was determined by auscultation of the lungs to determine the position of the catheter, and the respiratory sounds of the sides were symmetrically clear, so that the catheter was fixed and mechanical ventilation was performed. Anesthesia was maintained with remifentanil 0.1～0.3μg/(kg-min), propofol 2~4mg/(kg-h) rate microinfusion pump for continuous infusion. BIS was kept between 40~60. Intraoperative rocuronium bromide was given intermittently to maintain muscle relaxation. Perioperative fluid replacement followed the (4:2:1) rule in all patients. For maintenance of hemodynamic stability, ephedrine or atropine was administered, at the anesthesiologist's discretion, if verified a

SUMMARY:
Patients were randomly assigned to the GA group, PECS II group, or TPVB group using a computer-generated random number table. Group assignments were kept in a sealed envelope, which was opened only after induction of general anesthesia on the day of surgery. This study was a double-blind trial, ensuring that neither the patients nor the investigators were aware of the analgesic method used. The same anesthesiologist was responsible for PECS II block or TPVB, while different anesthesiologists were responsible for anesthesia implementation and postoperative follow-up.

DETAILED DESCRIPTION:
Written informed consent was obtained from all participants.90 female patients aged 18 to 65 with ASA I-II status were selected at Baogang Hospital, Inner Mongolia, who had been diagnosed with breast fibroadenomas. Exclusion criteria included pre-existing infection at the site of block, coagulation disorders, morbid obesity (body mass index > 40 kg/m²), allergy to local anesthetics, impaired lung function, significant cardiac disease, renal dysfunction, pre-existing neurological disorders, and psychiatric conditions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast fibromas

Exclusion Criteria:

* heart attack mental disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in visual analog scale scores | From enrollment to the end of treatment at 1 week
  Zero is equivalent to no pain and 10 indicates the worst possible pain."

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No
Research data is not shared for the protection of subjects